CLINICAL TRIAL: NCT07098676
Title: Haemodialysis Alters Hypercoagulability of Blood in Dialysis Patients
Acronym: TAT-t-PAIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: TAT-t-PAIC; SHYS-IEC-5.0/22K162/P01 (Registry Identifier: SHYS-IEC-5.0/22K162/P01)
Record Dates: First submitted 2025-06-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Individuals (Controls); Vascular Surgery Patients With Acute Thrombosis; Dialysis Patients
Keywords: thrombin-thrombomodulin complex (TM); thrombin-antithrombin complex (TAT); plasmin-α2-plasmin inhibitor complex (PIC); tissue plasminogen activator-inhibitor complex (t-PAIC); TAT/PIC ratio; diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteer: (1) aged between 18 and 85 years; (2) without any clinically diagnostic severe diseases including but not limited to a tumor, diabetes, cardiovascular, renal, nervous, digestive and mental disorders
- Vascular surgery patients with acute thrombosis: Inclusion criteria (1) Confirmed Imaging Evidence: Definitive visualization of a thrombus using imaging modalities such as ultrasonography (e.g., Doppler ultrasound for deep vein thrombosis), computed tomography (CT) pulmonary angiography, or magnetic resonance imaging (MRI) venography. (2) Consistent Clinical Presentation Supported by Imaging: A clinical picture suggestive of thrombosis (e.g., limb swelling, pain, or respiratory distress) corroborated by positive imaging findings. (3) Laboratory and Clinical Correlation: Elevated levels of a laboratory marker, such as D-dimer, combined with imaging evidence of thrombosis, and exclusion of alternative causes of symptoms (e.g., conditions listed in pregnancy registries or other differential diagnoses). Exclusion criteria were: (1) blood samples collected more than 24 hours after the thrombotic event; (2) blood samples taken while patients were using small-molecule heparin or other medications that could alter blood coagulation status.
- Dialysis patients: The inclusion criteria included patients with end-stage chronic kidney disease (eGFR≤15 mL/(min·1.73m²)) who had been on regular dialysis at the hospital for at least three months. Exclusion criteria were: (1) hemodialysis patients with no recent history of major surgical conditions or other diseases that could influence hemagglutination; (2) patients not on regular dialysis for at least three months; (3) patients who did not provide informed consent or complete the Paruda scoring form.

SUMMARY:
Primary Objective:

To develop a thrombotic event risk assessment model integrating serum biomarkers (TM, TAT, t-PAIC, PIC) with clinical data, systematically compare its predictive performance across healthy populations, vascular surgery patients with acute thrombosis, and dialysis patients, and evaluate its predictive advantages over the Padua Prediction Score and D-dimer.

Secondary Objective:

To investigate the expression profiles of these four thrombotic biomarkers in different populations and their associations with thrombotic event types and clinical contexts (e.g., duration of dialysis, anticoagulation regimens), identifying independent risk factors and underlying mechanisms to provide a scientific foundation for stratified thrombotic risk management and personalized intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients: The inclusion criteria included patients with end-stage chronic kidney disease (eGFR≤15 mL/(min·1.73m²)) who had been on regular dialysis at the hospital for at least three months healthy volunteer：aged between 18 and 85 years; (2) without any clinically diagnostic severe diseases including but not limited to a tumor, diabetes, cardiovascular, renal, nervous, digestive and mental disorders Diagnostic Criteria for Thrombosis: (1) Confirmed Imaging Evidence: Definitive visualization of a thrombus using imaging modalities such as ultrasonography (e.g., Doppler ultrasound for deep vein thrombosis), computed tomography (CT) pulmonary angiography, or magnetic resonance imaging (MRI) venography. (2) Consistent Clinical Presentation Supported by Imaging: A clinical picture suggestive of thrombosis (e.g., limb swelling, pain, or respiratory distress) corroborated by positive imaging findings. (3) Laboratory and Clinical Correlation: Elevated levels of a laboratory marker, such as D-dimer, combined with imaging evidence of thrombosis, and exclusion of alternative causes of symptoms (e.g., conditions listed in pregnancy registries or other differential diagnoses).

Exclusion Criteria:

* dialysis patients: (1) hemodialysis patients with no recent history of major surgical conditions or other diseases that could influence hemagglutination; (2) patients not on regular dialysis for at least three months; (3) patients who did not provide informed consent or complete the Paruda scoring form.

Thrombosis: (1) blood samples collected more than 24 hours after the thrombotic event; (2) blood samples taken while patients were using small-molecule heparin or other medications that could alter blood coagulation status

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dialysis patients: The inclusion criteria included patients with end-stage chronic kidney disease (eGFR≤15 mL/(min·1.73m²)) who had been on regular dialysis at the hospital for at least three months Healthy volunteers Diagnostic Criteria for Thrombosis: (1) Confirmed Imaging Evidence; (2) Consistent Clinical Presentation Supported by Imaging: A clinical picture suggestive of thrombosis corroborated by positive imaging findings; (3) Laboratory and Clinical Correlation
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
thrombosis outcome in dialysis patients | 1 years
  1. Incidence of radiologically confirmed thrombosis Definition: Thrombus definitively visualized by ultrasonography, CT pulmonary angiography, or MRI venography.
  2. Incidence of clinically suspected thrombosis with imaging support Definition: Clinical presentation (e.g., limb swelling, pain, respiratory distress) with positive imaging findings.
  3. Incidence of laboratory-supported thrombosis with imaging evidence Definition: Elevated D-dimer levels + positive imaging findings + exclusion of alternative diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Changbin Li, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No